CLINICAL TRIAL: NCT00352664
Title: Donepezil for Cancer Patients With Sedation Related to Opioid Treatment: A Double-blind Placebo Controlled Randomized Study
Brief Title: The Effect of Donepezil on Sedation and Other Symptoms
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low patient accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Eduardo Bruera, MD / Professor, UT MD Anderson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2003-0425
Record Dates: First submitted 2006-07-12; First posted 2006-07-14 (Estimated); Results first posted 2009-12-29 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2009-12

CONDITIONS: Advanced Cancer
Keywords: Advanced Cancer; Cancer Pain; Donepezil; Sedation; Placebo
MeSH Terms: conditions — Cancer Pain | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Donepezil (Active Comparator): Oral Donepezil 5 mg daily x 7 days
  Interventions: Drug: Donepezil
- daily x 7 days (Placebo Comparator): Placebo tablet daily x 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Donepezil — 5 mg once a day by mouth for 7 day cycle. After evaluation on Day 8, all participants will be offered donepezil every day for 7 days.
  Other Names: Aricept
  Arms: Donepezil
Drug: Placebo — Placebo tablet once a day by mouth for one 7 day cycle. After evaluation on day 8, all participants offered donepezil every day for 7 days.
  Arms: daily x 7 days

SUMMARY:
Primary Objective:

1. To determine the effectiveness of donepezil as compared to placebo for the management of opiate-induced sedation/drowsiness in patients with stable cancer pain

Secondary Objectives:

1. To assess the side-effects in both groups of 1 week treatment of 5 mg donepezil and placebo
2. To assess the effects of donepezil on fatigue (FACIT-Fatigue), and other symptoms (Anderson Symptom Assessment Scale)
3. To assess the effects of donepezil on cognition (Symbol Digit Modalities Test)
4. To assess the effects of donepezil on constipation (number of bowel movements)

DETAILED DESCRIPTION:
Donepezil is currently used in the treatment of certain types of mental disorders, including Alzheimer's disease. Recent research studies have shown that donepezil helps to improve drowsiness in cancer patients receiving opioid medication.

Before treatment starts, you will be asked to answer some questions regarding your cancer diagnosis, the medication you are taking, and the symptoms you are having (i.e. pain, fatigue, nausea, depression, anxiety, drowsiness, shortness of breath, appetite, sleep problem, constipation, and well-being) and a test for your cognitive status (matching specific numbers with given geometric figures) will be performed. It will take about 30 minutes to complete the evaluation. Women who are at risk of being pregnant must have a negative urine pregnancy test.

If you are qualified to enter the study you will be randomly assigned (as in the toss of a coin) to one of two groups. Participants in one group will receive donepezil for one week. Participants in the other group will receive a placebo (a tablet that does not contain any medication but looks just like the donepezil pill). You will have an equal chance (50/50) of being placed in either group. Neither you nor any the medical staff or researchers on this study will know if you are receiving the study drug or the placebo.

You will take 1 tablet of donepezil/placebo a day for 7 days. The research nurse will contact you by phone (in person if you are in the hospital) daily to ask questions about side effects and other symptoms.

On Day 8, you will need to come to the palliative care clinic for an evaluation. If you can not come to clinic on day 8, evaluation will be performed through telephone. Evaluation of sedation/drowsiness, pain, constipation, fatigue, side effects, effectiveness of the treatment, and a test of nervous system and cognitive status will be performed. If you develop intolerable side effects while on this study, the medication will be stopped and you will be removed from the study.

After evaluation on Day 8, all participants will be offered the chance to receive 1 tablet of donepezil every day for 7 days. The research nurse will follow up with you by phone (in person if you are in the hospital) 3 or 4 days after you received donepezil (open label) to ask questions about side effects and other symptoms.

On Day 15, you will need to come to the palliative care clinic for an evaluation. Evaluation of sedation/drowsiness, pain, constipation, fatigue, side effects, effectiveness of the treatment, and a test of nervous system and cognitive status will be performed. You will be given an option to continue on an additional 8 weeks. During these 8 weeks, the follow up will be conducted by your primary physician.

This is an investigational study. Donepezil has been approved by FDA and is a commercially available drug. Its use in this study is investigational. It can continue to be prescribed by your primary physician after that time if needed. A total of 100 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with drowsiness/sedation caused by opiate for > 3 days and its intensity more or equal to 3/10 (0 to 10 scale; 0 = no sedation, 10=worst possible sedation).
2. Patient receiving a regular dose of a strong opioid for the treatment of cancer pain, and no dose changes or dose change within 50% for at least 48 hours.Regular administration, defined as short acting opioids oral or parenteral every 4 hours around clock, slow release oral opioids every 12 hs or 24 hs, or transdermal opioids every 72 hours. Strong opioids include morphine, hydromorphone, methadone, fentanyl, and oxycodone.
3. Patient with relatively intact cognition defined by the Mini Mental State Examination according to age and educational level. A score of 24 or above is usually considered normal.
4. Patient willing to engage in follow up visit with a nurse by phone on day 2-7 (each day), 11 and 15 of the study and to return for follow up visit on day 8 of treatment. If patient is unable to come to clinic, assessment will be performed through telephone.
5. Sexually active females at risk of being pregnant with a negative urine pregnancy test
6. Written consent form signed.
7. Patients are 18 years or older
8. Concurrent radiation treatment (defined as 10 or less fractions for a palliative indication) is allowed
9. Concurrent chemotherapy is allowed, if the first two cycles have been well tolerated (defined as no grade 3 or 4 non-hematological toxicity)

Exclusion Criteria:

1. Major contraindication to donepezil i.e. hypersensitivity to donepezil or piperidine derivatives.
2. Patients in whom a major change in opiate dose, analgesia requirements, anesthetic procedures or general anesthetic is expected over the next seven days.
3. Treatment with anti-cholinergic agents (i.e., glycopyrrolate)
4. Patients taking Methylphenidate.
5. Patients with tube feeding (due to difficulty of accurate assessing some of the symptoms such as appetite and anorexia).
6. History of ongoing arrhythmia causing a rhythm other than a sinus rhythm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2003-11; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Bruera, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T. M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient Recruitment: 12/10/03 for first patient through 09/14/05 for last patient. All participants recruited at UT MD Anderson Cancer Center.
Pre-assignment Details: 27 patients were enrolled, 7 dropped out prior to assessment and were excluded from the overall study. Due to early termination, patients were not randomized.
Groups:
- Placebo: Oral Placebo tablet daily x 7 days
Period: Overall Study
Arm/Group | Donepezil | Placebo
Started | 27 | 0
Completed | 20 | 0
Not Completed | 7 | 0
Not completed — Withdrawal by Subject | 7 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Donepezil | Placebo | Total
Number analyzed (Participants) | 27 | 0 | 27
Age, Continuous [Median (Full Range); unit: years] | 56 [22 to 64] |  | 56 [22 to 64]
Gender [Number; unit: participants]
  Female | 18 |  | 18
  Male | 9 |  | 9
Region of Enrollment [Number; unit: participants]
  United States | 27 |  | 27

OUTCOME MEASURES:

1. Primary Outcome: Sedation Mean Scores at 1-Week
Description: Anderson Symptom Assessment Scale (ASAS) was used to measure sedation mean scores (SD) on a 0-10 scale with 0 representing "not drowsy" and 10 representing "worst possible drowsiness."
Time Frame: Baseline and Day 7
Population: Analysis was intention to treat (ITT), and population analyzed was that treated. Study closed early due to low patient accrual and insufficient supply of drug. No patients were randomized to Placebo Arm.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 20 | 0
Scores on a Scale
  Baseline | 6.44 (1.2) |
  Day 7 | 4.81 (2.6) |

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Donepezil | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/0
Other Adverse Events (participants affected / at risk) | 17/20 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Donepezil (N=20) | Placebo (N=0)
Nausea/vomiting (Gastrointestinal disorders) | 6 (6) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 0 (0)
Anorexia (General disorders) | 4 (4) | 0 (0)
Muscle Cramps (General disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Insufficient drug supply and low patient accrual closed study early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No